CLINICAL TRIAL: NCT02624999
Title: An Individualized Cancer Vaccine for Recurrent/Metastatic (R/M) Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Study Comparing AlloVax™ to Chemotherapy in Recurrent/Metastatic Squamous Cell Carcinoma of the Head & Neck
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI changed institution
Sponsor: Mirror Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITL-020-HENK-VAXPII
Record Dates: First submitted 2015-11-29; First posted 2015-12-09 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2016-07

CONDITIONS: Squamous Cell Carcinoma Head and Neck
Keywords: Head and Neck Cancer; SCCHN; R/M SCCHN; Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Carcinoma | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immunotherapy (Experimental): Subjects in this arm will receive immunotherapy (AlloVax™: CRCL + AlloStim™) twice a week for 4 weeks and then every 4 weeks for an additional 12 weeks
  Interventions: Biological: AlloVax™
- Standard chemotherapy (Active Comparator): Subjects in this arm will receive up to six three-week cycles of chemotherapy consisting of cisplatin on day 0 of the 3-week cycle at dose 80-100 mg/m2 IV followed by 1000 mg/m2 IV 5FU on days 1-4 of the cycle
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Biological: AlloVax™ — AlloVax™ combines an anti-tumor effect of mini-transplant procedures with patient specific tumor antigens
  Other Names: CRCL + AlloStim™
  Arms: Immunotherapy
Drug: Cisplatin — Subjects in the chemotherapy arm will receive up to 6 cycles of cisplatin on day 0 of the 3-week cycle at dose of 80-100 mg/m2 IV and 1000 mg/m2 IV 5FU on days 1-4 of the cycle
  Other Names: Standard Chemotherapy
  Arms: Standard chemotherapy

SUMMARY:
Phase II, Randomized, Non-Inferiority Study Comparing an Individualized Cancer Vaccine (AlloVax™) to Chemotherapy in Subjects with R/M SCCHN .

DETAILED DESCRIPTION:
All accrued subjects will be randomized 2:1 to AlloVax™ (CRCL + AlloStim™) immunotherapy vs. standard chemotherapy. AlloVax™ is an experimental individualized therapeutic vaccine shown to be active in this study population.

The standard chemotherapy arm (Arm 1) will receive up to six three-week cycles of chemotherapy consisting of cisplatin on day 0 of the 3-week cycle at dose 80-100 mg/m2 IV followed by 1000 mg/m2 IV flurouracil (5FU) on days 1-4 of the cycle.

The immunotherapy arm (Arm 2) will receive immunotherapy (AlloVax™) twice a week for 4 weeks and then every 4 weeks for an additional 12 weeks.

The study is designed and powered to determine if AlloVax™ is not inferior to the active chemotherapy control.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and female subjects aged 18 years or older at screening visit.
* Histopatholologically or cytologically confirmed diagnosis of locoregionally recurrent unresectable or previously untreated metastatic SCCHN.
* Tumor lesion safely accessible for biopsy or surgical excision resulting in a minimum of 0.2 g of tumor sample for CRCL processing.
* Subjects must have measurable disease according to revised RECIST v.1.1 guidelines.
* Eastern Cooperative Oncology Group (ECOG) ≤1.
* Subjects must be screened to be negative for Human Immunodeficiency Virus 1 (HIV1), HBsAg, Hepatitis C (HCV) and Rapid Plasma Reagin (RPR,syphilis).
* Subjects must have adequate organ function including: (WBC >3000/mm3, Platelets >100,000/mm3, Absolute neutrophil count ≥ 1,500/mm³, Hemoglobin ≥ 10.0 g/dL (transfusion allowed)), Hepatic (Serum Total bilirubin < 2 x ULN mg/dL, Alanine transaminase (ALT) (SGPT) / Aspartate aminotransferase (AST) (SGOT) ≤3 x upper limit of normal (ULN)), Renal: Serum creatinine (SCR) <2.0 x ULN, or, Creatinine clearance (CCR) >30 mL/min.
* Pre-study EKG without significant abnormalities.
* Women of child-bearing potential must have a negative urine or serum pregnancy test result within 72 hours prior to the start of study drug administration.
* If child producing potential age, must agree to use contraception or avoidance of pregnancy measures while enrolled on study and receiving the experimental product.
* Ability to understand the study, its inherent risks, side effects and potential benefits and be able to give written informed consent to participate.

Exclusion Criteria:

* Clinical evidence or radiological evidence of brain metastasis.
* Treated for another primary cancer within 2 years prior to signing inform consent form.
* Any concomitant anticancer therapies.
* History of severe hypersensitivity to monoclonal antibody drugs or any contraindication to any of the study drugs.
* Concomitant active autoimmune disease (e.g., rheumatoid arthritis, multiple sclerosis, autoimmune thyroid disease, uveitis).
* Prior experimental therapy or cancer vaccine treatment (e.g., dendritic cell therapy, heat shock vaccine).
* Clinical requirement for systemic steroids or immunosuppressive therapy, including: cyclosporine, antithymocyte globulin, or tacrolimus within 1 month prior to signing inform consent form.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, requiring parenteral antibiotics, symptomatic congestive heart failure, severe myocardial insufficiency, cardiac arrhythmia. All infections must be resolved and the subject must remain a febrile for seven days prior to being placed in the study.
* History of blood transfusion reactions.
* Psychiatric or addictive disorders or other condition that, in the opinion of the investigator, would preclude study participation.
* Female subject is pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Estimated); Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (vital signs, physical examination, clinical laboratory profile, adverse events assessed by CTCAE v4.0 and dose limiting toxicity (DLT)) | 119 days
  Whether AlloVax™ is less toxic than chemotherapy. will be evaluated on the basis of the following parameters: vital signs, physical examination, clinical laboratory profile, adverse events assessed by CTCAE v4.0 and dose limiting toxicity (DLT)
Overall Survival | 119 days
  Whether AlloVax™ is not inferior to the active chemotherapy control (from time of randomization). Subjects are followed for survival during the trial and as long as they are alive after the last study treatment through follow-up

SECONDARY OUTCOMES:
Health related Quality of Life (HRQoL) | 119 days
  QLQ-C30 and QLQ-H&N35 questionnaires

OTHER OUTCOMES:
RECIST | 119 days
  Response and correlation with pathology assessment
Immune-Related Response Criteria (irRC) | 119 days
  Response and correlation with pathology assessment
Immune response in the treatment arm | 119 days
  Correlation of OS with immune response

CONTACTS AND LOCATIONS:
Overall Officials: Michael Har-Noy, Dr., Study Director — CEO & CTO
Locations (1):
- National Cancer Institute of Thailand, Bangkok, Thailand